CLINICAL TRIAL: NCT06337786
Title: A Randomized Controlled Clinical Trial Investigating the Effects of the Digital App Rheumabuddy4.1 in Patients With Rheumatoid Arthritis
Brief Title: Investigating the Effects of the Digital App Rheumabuddy4.1 in a Clinical RCT Set-up in Patients With Rheumatoid Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henning Bliddal (Other)
Collaborators: Eurostars (Other); DAMAN (Unknown); Medical University of Vienna (Other)
Responsible Party: Sponsor-Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MSK-2023-TSJ1
Record Dates: First submitted 2024-03-14; First posted 2024-03-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Patient Perspectives; Digital app; Quality of life; Empowerment; Socioeconomic burden
MeSH Terms: conditions — Arthritis, Rheumatoid; Empowerment

STUDY DESIGN:
Intervention Model Description: The trial is an open-label randomized controlled clinical trial with two parallel groups .
  The participants will be randomly allocated in a 1:1 manner receiving either standard care and the digital app RB4.1 or standard care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Patients diagnosed with rheumatoid arthritis receiving standard care and the digital app RB4.1
  Interventions: Device: Digital app RB4.1
- Control arm (Active Comparator): Patients diagnosed with rheumatoid arthritis receiving standard care alone.
  Interventions: Other: Control arm

INTERVENTIONS:
Device: Digital app RB4.1 — Standard care and the digital app RB4.1
  Arms: Intervention arm
Other: Control arm — Standard care alone
  Arms: Control arm

SUMMARY:
Rheumatoid arthritis (RA) is one of the most frequently occurring autoimmune rheumatic diseases, affecting an estimated 1% of the global population. RA is a chronic inflammatory disease that leads to the development of synovial inflammation and effusion, ultimately followed by joint destruction and permanent disability.

The substantial socioeconomic burden and the challenge of RA patients adhering to treatment is an important factor of this disease and its impact on both patients and society. An innovative approach is needed in order to find new ways to assist and truly empower patients to understand their disease, increase compliance and thereby increase quality of life.

There is a discrepancy in the understanding of what's of importance when living a life with a chronic disease. The importance of patients' perspectives concerning disease- and treatment related impacts, is of crucial importance when involving patients in decisions about treatment, and to support the patients in optimal medication-taking behaviour to ensure patient health and reduce health care costs. There are still unmet needs that have a huge impact on quality of life (QoL) such as fatigue, pain, sleep and psychological issues, etc, which need to be taken seriously as these can have severe and debilitating consequences for the individual.

The aim of this study is to investigate and evaluate the effects of the digital app RheumaBuddy4.1 (RB4.1) and the ability to provide support and increase quality of life in patients with RA

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) incurs a substantial socioeconomic burden which has been supported by the Global Burden of Disease studies. The substantial socioeconomic burden and the challenge of RA patients adhering to treatment is an important factor of this disease and its impact on both patients and society.

An innovative approach is needed in order to find new ways to assist and truly empower patients to understand their disease, increase compliance and thereby increase quality of life.

Many RA patients experience a gap between the health care professionals (HCPs) and the patients regarding the understanding of living a life with a chronic disease - it is more than just blodsamples and swollen/tender joints.This trial addresses a critical, previously not well addressed, question of patient- and clinical importance about the support of using electronically patient reported outcomes (ePROs) ensuring high-quality life living with a chronic disease in patients with RA.

Digital health technology, as adjunct to standard routine care, provides a big opportunity to deliver continuous relevant, timely and cost-effective support to patients including support behavioural changes, improve quality of life and optimize treatment. Many (86%) of patients with RA agree that RA self-management apps can be very helpful, but the lack of high-quality and scientifically validated apps are needed.

The trial will create an evidence base covering the implications of disease- and treatment related concerns as well as non-adherence on quality of life (QoL), patient empowerment, clinical symptoms, and use of medication. Decision and policy makers need a transparent evidence base to substantiate the judgment behind any rational clinical rheumatology practice. The methodology is based on a 'bottom up' approach that hopefully will provide a state-of-the-art model for ensuring patient value in health care settings.

Altogether it is very likely that the use of data collected in RB4.1 will be of significant benefit to both patients with RA and HCPs.

The aim of this study is to investigate and evaluate the effects of the digital app RheumaBuddy4.1 (RB4.1) and the ability to provide support and increase quality of life in patients with RA

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all of the following criteria to be enrolled in the study:

1. Diagnosed with RA according to the EULAR & American College of Rheumatology
2. PGA level >= 40mm
3. Age ≥ 18 years and < 65 years
4. Motivated for the intervention
5. Willing and able to understand and participate in the study
6. DAS28-CRP ≤ 3.2.
7. Ability to use the RB4.1 app

Exclusion Criteria:

An individual will be excluded from the study if she meets any of the following criteria:

1. Dementia or other linguistic/cognitive/physical deficiency that prevents participation
2. Vision impairment that prevents the use of the devices and computer
3. Change in DMARD (within 8 weeks)
4. Chronic widespread pain (fibromyalgia) based on patient anamnesis/medical record.
5. Acute infections based on patient anamnesis/medical record.
6. Severe asthma based on patient anamnesis/medical record.
7. Severe COPD based on patient anamnesis/medical record.
8. Instable heart disease based on patient anamnesis/medical record.
9. Intensive physiotherapy outside standard care based on patient anamnesis/medical record.
10. Electrostimulation based on patient anamnesis/medical record.
11. Motivation training based on patient anamnesis/medical record.
12. Smoking based on patient anamnesis/medical record.
13. Fever based on patient anamnesis/medical record.
14. If pain/fatigue are considered a side effect judged by the treating physician.
15. Other autoimmune diseases based on patient anamnesis/medical journal.
16. Mental diseases based on patient anamnesis/medical record.
17. All other non-pharmacological therapies that may impact the course of RA judged by the treating physician.
18. Any comorbid condition, that in the opinion of the investigator would interfere with the conduction of the trial or the interpretation of the study outcome.
19. Previous use of health apps related to the RA disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patient Global Assessment | Week 12, Week 24, change from baseline
  Patient Global Assessment (PGA) is scored using a visual analogue scale (VAS) range from 0-100 mm. Higher scores represent a higher level of disease activity or a worse global health.
  The PGA is one of the most widely reported PROs in RA. The considerable burden of RA on the individual is related to both inflammation and damage but also to broader aspects of disease, including psychological and societal impact. The way PGA is used in clinical practices covers, in fact, two very different concepts, one related to global health and the other to overall disease activity They are both usually used under the heading of PGA without further specification for which is being assessed.

SECONDARY OUTCOMES:
Disease-activity Score28 using C-reactive protein (DAS28-CRP) | Week 12, Week 24, change from baseline
  Disease activity of rheumatoid arthritis (RA) is usually assessed by using Disease Activity Score 28-joint count (DAS28). DAS28 is a validated composite measure combining patient-reported outcomes and clinical measures of inflammation and has been widely adopted in RA trials and clinical practice, providing a robust measure for assessing intervention efficacy. DAS28 scores range from 0 to 9.4 and are calculated using tender joints, swollen joints, general health, and a laboratory measure of acute inflammation. DAS28 for RA with C-reactive protein (DAS28-CRP) describes the severity of RA using clinical and laboratory data, specifically CRP.
Self-Efficacy (ASES-8) | Week 12, Week 24, change from baseline
  The ASES was developed to measure patients 'arthritis-speciﬁc self-efﬁcacy, or patients' beliefs that they could perform speciﬁc tasks or behaviors to cope with the consequences of arthritis. ASES-8 has been used in evaluations of self-management education programs, physical activity interventions, and associations of self-efficacy with various health outcomes. The ASES-8 includes 2 items from the ASES pain subscale, 4 items from the ASES other symptoms subscale, and 2 new items related to preventing pain and fatigue from interfering with things you want to do. The total scale includes 8 items with no subscales: 1 (very uncertain) to 10 (very certain). Item stem for each question begins "How certain that you can....". The score for the scale is the mean of the eight items.
Pain (VAS) | Week 12, Week 24, change from baseline
  Pain are the most common and debilitating symptoms of RA, significantly impacting patients' quality of life. Pain will be assessed using the 0-100 mm visual analogue scale (VAS) with anchors 0 = "no pain" and 100 = "Worst imaginable pain".
Fatigue (VAS) | Week 12, Week 24, change from baseline
  Fatigue is a very common and debilitating symptoms of RA, significantly impacting patients' quality of life. Fatigue will be assessed using the 100 mm visual analogue scale (VAS) with anchors 0 = "no fatigue" and 100 = "Worst imaginable fatigue".
Health related quality of life (EQ-5D) | Week 12, Week 24, change from baseline
  The EQ-5D questionnaire is developed by the EuroQoL. The EQ-5D is a five-dimensional health state classification. The five dimensions are mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It is a preference-based measure that can be regarded as a continuous outcome scored on a -0.59 to 1.00 scale, with 1.00 indicating 'full health' and 0 representing dead. The negative EQ-5D scores represent certain health states valued as worse than dead. Each topic is rated on a 3-point Likert scale: 1) no problems, 2) some problems, and 3) extreme problems. Instructions on how to response is included in the questionnaire. In addition, a VAS scale functions as a 6-question to report on self-reported overall health on a 0-100 scale where 100= best imaginable health and 0=worst health you can imagine. The VAS can be used as a quantitative measure of the patient's own judgement of overall health.
Physical function (MD-HAQ) | Week 12, Week 24, change from baseline
  The Multi-Dimensional Health Assessment Questionnaire (MD-HAQ) is derived from the HAQ Health Assessment Questionnaire, which includes an index of the three rheumatoid arthritis (RA) core data set measures (physical function, pain and global estimate). It consists of 10 questions addressing eight different areas of functional ability and yields a total score between 0 and 3, with a higher score representing increasing disability. The MD-HAQ is useful in all rheumatic diseases by saving time, documenting changes in status over long periods and by improving rheumatology care and outcomes.
Well-Being (WHO-5) | Week 12, Week 24, change from baseline
  Mental health is a state of mental well-being that enables people to cope with the stresses of life, realize their abilities, learn well and work well, and contribute to their community. Well-Being will be assessed using the 5-item Well-Being Index (WHO-5). The WHO-5 is a validated assessment tool used to measure mental well-being in a variety of patient populations. The raw score is calculated by totalling the figures of the five answers. The raw score ranges from 0 to 25; 0 representing worst possible quality of life and 25 representing best possible quality of life.
Medication Adherence (MMAS-8) | Week 12, Week 24, change from baseline
  Adherence to medication will be assessed using the 8-item Morisky Medication Adherence Scale (MMAS-8). The MMAS-8 is a validated assessment tool used to measure non-adherence in a variety of patient populations. The scale consists of eight questions, MMAS-8 scores can range from 0 to 8 points. According to the MMAS-8, adherence can be categorized as high adherence (score, 8), medium adherence (score, 6 to<8) and low adherence (score, <6).
Perceived Efficacy in Patient-Physician Interactions (PEPPI-5) | Week 12, Week 24, change from baseline
  The Perceived Efficacy in Patient-Physician Interactions (PEPPI) scale was developed to measure older patients' self-efficacy in both obtaining medical information and attention to their chief health concern from a physician. The PEPPI 5-item short form will be used to assess adherence and was developed from the items demonstrating the most variability while maintaining adequate internal consistency and construct validity from the original PEPPI. The PEPPI-5 includes five items; each item starts with "how confident are you in your ability to..? " Items are rated by participants from one to five; 1 = "not at all confident",5= "very confident". The totalled results are in the range of 5 to 25; higher scores indicate that the participant has higher self-efficacy in patient-physician interactions .

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, Principal Investigator — The Parker Institute, Bispebjerg and Frederiksberg Hospital
Locations (1):
- The Parker Institute, Bispebjerg and Frederiksberg Hospital, Frederiksberg, Copenhagen F, Denmark